CLINICAL TRIAL: NCT06376734
Title: Transdiagnostic Circuit Mapping of Prefrontal Targets in Accelerated Transcranial Magnetic Stimulation
Brief Title: Search for Novel Transcranial Magnetic Stimulation (TMS) Targets for Mental Illness
Acronym: Expedition
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Shan Siddiqi, MD, Principal Investigator, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2024p000528
Record Dates: First submitted 2024-03-31; First posted 2024-04-19 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder; Obsessive-Compulsive Disorder; Schizophrenia; Generalized Anxiety Disorder; Mood Disorders; Psychiatric Disorder; Mental Disorder; Depression, Anxiety
Keywords: depression; anxiety; schizophrenia; OCD; obsessive-compulsive disorder; transcranial magnetic stimulation; TMS; accelerated TMS; accelerated intermittent theta burst stimulation; brain stimulation; neuromodulation; transdiagnostic; neuronavigation; functional connectivity; neuroimaging; theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Obsessive-Compulsive Disorder; Schizophrenia; Generalized Anxiety Disorder; Mood Disorders; Mental Disorders; Depression; Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled crossover trial. Participants will be stimulated at a random location in the prefrontal cortex, which will be mapped to its underlying brain network to determine which network was stimulated.
Masking Description: All participants will receive real open-label TMS, so there will be no conventional masking. However, participants and investigators will be blinded to which network is being stimulated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TMS to random PFC location 1 (Experimental): Participants will receive 2 days of accelerated TMS (10 treatments per day) to a random location in the prefrontal cortex.
  Interventions: Device: Transcranial magnetic stimulation
- TMS to random PFC location 2 (Experimental): After a 2-month washout following arm 1, participants will receive another two days of accelerated iTBS treatment at a different random PFC location.
  Interventions: Device: Transcranial magnetic stimulation
- TMS to Schizophrenia location (Experimental): Patients with schizophrenia will be offered to participate in a third arm of the trial, during which participants will receive 2 days of accelerated iTBS to a schizophrenia-specific target.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Accelerated TMS will be provided for 2 days using the same dosing regimen as the FDA-cleared SAINT protocol, ten 9-minute treatments per day.

SUMMARY:
Participants will receive Transcranial Magnetic Stimulation (TMS) at a random location in the left prefrontal cortex, excluding sites that are potentially unsafe. Extensive behavioral testing will be conducted to determine which behaviors are modulated by stimulating which circuits.

DETAILED DESCRIPTION:
Patients who meet inclusion criteria for a primary diagnosis of MDD, OCD, GAD, or Schizophrenia (n=90) and consent to treatment will be assigned two random stimulation sites in the left prefrontal cortex and receive 2 days of accelerated iTBS treatment at the first stimulation site. Patients will have a 2 month break before coming back for 2 days of accelerated iTBS treatment at the second stimulation site. Patients with schizophrenia will be offered to participate in a third arm of the trial using a schizophrenia-specific target. This arm will also include fMRI scans and behavioral testing pre- and post- aiTBS. There will be two days (6 hours total) of behavioral testing and MRI scanning before each stimulation session and two days (6 hours total) after each stimulation session. Participants will be given the option of completing the behavioral testing in one day, before and after stimulation sessions. All the patients will receive active stimulation, which will facilitate enrollment and eliminate ethical concerns about placebo treatment in vulnerable patient populations. All participants will be blinded to their target coordinates and scales will be administered by a blinded study staff.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* English proficiency sufficient for informed consent, questionnaires/tasks, and treatment
* Primary diagnosis of one of the following: major depressive disorder (MDD), obsessive-compulsive disorder (OCD), generalized anxiety disorder (GAD), or schizophrenia (determined by focal assessment using the Structured Clinical Interview for DSM-5)

  * ≥20 on the Beck Depression Inventory for patients with MDD
  * ≥16 on the Beck Anxiety Inventory for patients with GAD
  * ≥16 on the Yale-Brown Obsessive-Compulsive Scale for patients with OCD
  * ≥58 on the Positive and Negative Symptom Scale for patients with schizophrenia
* Stable psychotropic medication regimen, or remain medication free, for 4 weeks prior to treatment (Medication changes during study enrollment period will be tracked for post hoc analysis).
* Primary clinician (e.g. psychiatrist, therapist, psychologist, APRN, PA, etc.) responsible for psychiatric care before, during, and after the trial

Exclusion Criteria:

* Active pregnancy as determined by a urine pregnancy test
* Cluster B personality disorders (antisocial personality disorder, borderline personality disorder, histrionic personality disorder, narcissistic personality disorder)
* PTSD with active, clinically significant symptoms, as determined by clinician
* Diagnosis of Schizoaffective Disorder, Bipolar Type
* Recent (within 4 weeks) or concurrent use of rapid-acting antidepressant agent (ketamine/esketamine/ECT)
* Ferromagnetic metallic implant that would contraindicate receiving TMS or obtaining MRI
* Any other TMS or MRI safety concerns identified by the clinician
* Receiving or planning to receive other TMS treatments during course of participation
* History of:

  * Neurosurgical intervention for mental illness
  * Moderate to severe autism spectrum disorder
  * Intellectual disability
  * Severe cognitive impairment
  * Significant neurological illness (e.g., dementia, Parkinson's, Huntington's, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis)
  * Untreated or insufficiently treated endocrine disorder
  * Eating disorders
  * Treatment with investigational drug or intervention during the study period
* Current evidence of:

  * Mania or hypomania
  * Active suicidal ideation or a suicide attempt within the past year
  * Contraindications to either TMS or MRI (e.g., metallic implants, etc.).
  * Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
  * Significantly increased seizure risk as determined by a clinician
* For participants with schizophrenia:

  * Evidence of impaired capacity to consent, e.g. impaired insight into illness, as deemed by a licensed psychiatrist or psychologist on the study team
  * Hospitalization with psychosis in the past 6 months
* Positive urine drug screen for illicit substances
* Existing tinnitus (ringing in the ears)
* Any other condition deemed by the PI to interfere with the study or increase risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Clustering of multiple behavioral measures | through study completion, average of 3 months
  The primary outcome is that stimulation of different circuits will selectively modify different behavioral clusters. Participants will complete the following phenotyping battery tasks and questionnaires:
  Q-SCID PANSS SAPS SANS PYRATS CDSS YBOCS CGI ATQ ASI BAI BDI BIS/BAS Claremont Purpose Scale De Jong Gierveld Loneliness Scale Daily Spiritual Experience Scale Emotional Reactivity Scale Flourishing Measures Headache Impact Test HiTOP-Self Report Moral Judgment Scale Pain Screener Personal Relationship with God Scale PSQI Positive and Negative Affect Scale Ruminative Response Scale Self Compassion-Short Form Spiritual Transcendence Scale- Short Form Temporal Experience of Pleasure Scale Values and Beliefs of the American Public Altruistic Decision Task Balloon Analogue Risk Task DSIAT EEfRT MSIT ECR Time perception task TMB toolkit 5min AV recording

CONTACTS AND LOCATIONS:
Overall Officials: Shan H Siddiqi, MD, Principal Investigator — Brigham and Women's
Locations (2):
- United States (2):
  - Acacia Clinics, Sunnyvale, California
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
De-identified survey response data and/or neuroimaging data may be shared with collaborators for further analysis.